CLINICAL TRIAL: NCT05877885
Title: Targeting Network Dysfunction in Apathy of Late-life Depression Using Digital Therapeutics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-09025304; K23MH129882 (NIH)
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Major Depressive Disorder; Apathy
MeSH Terms: conditions — Depressive Disorder, Major; Lethargy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Cognitive Training Intervention (Experimental)
  Interventions: Behavioral: Targeted Cognitive Training Intervention
- General Cognitive Training Intervention (Active Comparator)
  Interventions: Behavioral: General Cognitive Training Intervention

INTERVENTIONS:
Behavioral: Targeted Cognitive Training Intervention — In this intervention, participants will complete 25-30 minutes of cognitive training per day, 5 days/week (but up to 7 days/week) for 4 weeks. The training protocol will be delivered via the Posit Science Platform, and includes tasks that emphasize training of sustained attention, salience detection, and dimensions of cognitive control. During the 4 week intervention, participants will have weekly 10-20 minute visits with a Care Manager to provide clinical monitoring of symptoms and structured support to participants.
  Arms: Targeted Cognitive Training Intervention
Behavioral: General Cognitive Training Intervention — In this intervention, participants will complete 25-30 minutes of cognitive activities per day, 5 days/week (but up to 7 days/week) for 4 weeks. The training protocol will be delivered via the Posit Science Platform. The intervention protocol will include computerized cognitive activities designed to provide general cognitive stimulation. During the 4 week intervention, participants will have weekly 10-20 minute visits with a Care Manager to provide clinical monitoring of symptoms and structured support to participants.
  Arms: General Cognitive Training Intervention

SUMMARY:
The goal of this randomized controlled trial is to evaluate the potential of a customized digital cognitive training intervention to target aspects of brain function in apathy of late-life depression and reduce symptoms of apathy and related cognitive and behavioral deficits. The investigators hypothesize that 4 weeks of a customized digital cognitive training program will lead to changes in brain connectivity, apathy severity, and cognitive control performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60+ years
2. Diagnosis of unipolar major depressive disorder without psychotic features, as assessed by the Mini International Neuropsychiatric Interview
3. Montgomery-Åsberg Depression Rating Scale (MADRS) score > or = 16.
4. Clinically significant apathy, determined by the Clinician-rated Apathy Evaluation Scale (C-AES > or = to 37)
5. Off antidepressants or on a stable dose of an antidepressant for 8 weeks and do not intend to change the dose in the next 5 weeks.
6. On a stable dose of other psychotropic medications, deemed by the investigator to be associated with brain networks of interest, for at least 8 weeks.
7. Capacity to provide written consent for research assessment and treatment
8. Ability to follow written and verbal instructions (English) as assessed by the PI and/or study staff.
9. Total score of > 29 on the Telephone Interview for Cognitive Status (TICS)
10. Eligible to undergo MRI
11. Access to a computer or tablet with Wifi capabilities
12. Able to comply with all testing and study requirements and willingness to participate in the full study duration.

Exclusion Criteria:

1. History or presence of psychiatric diagnoses other than major depressive disorder without psychotic features, persistent depressive disorder, generalized anxiety disorder, social anxiety disorder, or specific phobia
2. Use of cholinesterase inhibitors or psychoactive drugs other than antidepressants or benzodiazepines, including antipsychotics, that in the opinion of the Investigator may confound study data/assessments.
3. Presence or history of significant neurologic or neurodegenerative disorder (e.g., Alzheimer's disease and other dementias, amnestic Mild Cognitive Impairment, history of stroke, Multiple Sclerosis, Parkinson's disease, epilepsy).
4. Any other acute medical condition (e.g., cardiac, renal, or respiratory failure; severe chronic obstructive pulmonary disease; metastatic cancer; or debilitated states or less common medical illnesses) that may influence brain systems of interest or interfere with participation or interpretation of the study results.
5. Participant is currently considered at risk for attempting suicide by the Investigator, has made a suicide attempt within the past year, or is currently demonstrating active suicidal ideation or self-injurious behavior.
6. Electroconvulsive therapy within the past 12 months
7. Recent history (within 6 months prior to screening/baseline) of Substance Use Disorder.
8. Participant is currently enrolled in ongoing concurrent cognitive rehabilitation (note that if a subject is enrolled in psychotherapy, this will not be grounds for exclusion)
9. Claustrophobia
10. Color Blindness
11. Sensory or physical impairment that would preclude cognitive testing or participation in the intervention (e.g., upper limb paralysis) as reported by the participant or observed by the Investigator.
12. Travelling consecutively for 2+ weeks during the study period to a location that will preclude timely collection of post-treatment MRI data.
13. Contraindications to MRI scanning including cardiac pacemaker, heart valve replacement, vascular stent, cochlear implant, any other metallic biomedical implant contraindicating to MRI.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Resting State Functional Connectivity among the Salience, Executive Control, and Reward Networks | Baseline and Post-treatment (Week 4)
  Calculated from resting state fMRI scan. Validation of target engagement.

SECONDARY OUTCOMES:
Change in Apathy Evaluation Scale (AES) score | Baseline, Mid-treatment (Week 2), and Post-treatment (Week 4)
  The 18-item clinician-rated version of the Apathy Evaluation Scale (AES) will be used to measure apathy severity. Scores range from 18 (no apathy) to 72 (severe apathy).
Change in Stroop Interference score | Baseline, Mid-treatment (Week 2), and Post-treatment (Week 4)
  Stroop interference will be calculated from the computerized Stroop Task to measure cognitive control.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Oberlin, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Neuroscience Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared includes all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 3 months following publication of primary outcomes, ending 5 years following publication of primary outcomes.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal, to achieve the aims in the approved proposal. Proposals should be directed to the study PI, Lauren Oberlin, at lauren.oberlin@adventhealth.com